CLINICAL TRIAL: NCT07343843
Title: Effect of Virtual Reality Versus Intravenous Dexmedetomidine on Maternal Anxiety, Stress, Hemodynamics, and Neonatal Outcomes During Cesarean Section
Brief Title: Virtual Reality Versus Intravenous Dexmedetomidine on Maternal Anxiety, Stress, Hemodynamics, and Neonatal Outcomes During Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Emad Mohamed Sayed, Resident of Anesthesia and Intensive Care, Benha University, Benha, Egypt., Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.29.12.2025
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Virtual Reality; Dexmedetomidine; Maternal Anxiety; Stress; Hemodynamics; Neonatal Outcomes; Cesarean Section
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Following confirmation of adequate spinal anesthesia, dexmedetomidine will be administered as an intravenous infusion of 0.2-0.4µg/kg/hr until abdominal closure.
  Interventions: Drug: Dexmedetomidine
- Virtual reality group (Experimental): Participants will be fitted with virtual reality headsets immediately after the establishment of spinal anesthesia. The headsets will display calming immersive audiovisual content, and participants will continue wearing them throughout the entire procedure until skin closure.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Drug: Dexmedetomidine — Following confirmation of adequate spinal anesthesia, dexmedetomidine will be administered as an intravenous infusion of 0.2-0.4µg/kg/hr until abdominal closure.
  Arms: Dexmedetomidine group
Other: Virtual reality — Participants will be fitted with virtual reality headsets immediately after the establishment of spinal anesthesia. The headsets will display calming immersive audiovisual content, and participants will continue wearing them throughout the entire procedure until skin closure.
  Arms: Virtual reality group

SUMMARY:
This study aims to compare the efficacy of intravenous dexmedetomidine infusion versus virtual reality (VR) in reducing maternal anxiety, stress, and hemodynamic instability during cesarean section and their effects on neonatal outcome as respiration and heart rate.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most frequently performed surgical procedures worldwide, with steadily increasing rates across both developed and developing countries.

Dexmedetomidine, a highly selective α₂-adrenergic receptor agonist, has been increasingly utilized in obstetric anesthesia because of its anxiolytic, sedative, and analgesic properties with minimal respiratory depression.

Non-pharmacological interventions, such as virtual reality (VR), have emerged as innovative strategies for perioperative anxiety management. VR provides immersive distraction, thereby modulating pain perception and reducing stress.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* American Society of Anesthesiologists (ASA) physical status II.
* Scheduled for elective cesarean section (CS) delivery under Central Neuraxial Blockade.
* Provide informed consent and agree to participate in the study.

Exclusion Criteria:

* Patient's refusal
* Patient known have contraindications for Regional Anesthesia as infection at the site of injection, severe coagulopathy or allergy to local anesthetics.
* Patient with psychiatric disorders.
* Sensory impairment (blindness, deafness).
* Any technical problem preventing proper fitting of the glasses to the patient face.
* Patients with cognitive impairment, epilepsy or with claustrophobia
* Patients with suspected eye infection
* Signs of active labor.
* Pregnancy related-diseases or antepartum hemorrhage.
* Presence of Fetal distress.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women scheduled for elective cesarean section (CS) delivery.
Enrollment: 52 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maternal anxiety | Two hours postoperatively in the recovery room
  Maternal anxiety will be assessed at three time points (On admission to the operating theatre, At skin suturing, Two hours postoperatively in the recovery room) using the Novel Visual Facial Anxiety Scale (NVFAS), a validated pictorial self-report measure.
  NVFAS will be applied to measure acute state anxiety. This self-reported pictorial tool consists of 11 facial expressions corresponding to anxiety scores from 0 (no anxiety) to 10 (severe anxiety). The scale is user-friendly, language-independent, and has been validated for perioperative patients, including those with limited time for traditional questionnaires.

SECONDARY OUTCOMES:
Heart rate | 24 hours postoperatively
  Heart rate will be recorded at six predefined intra- and postoperative intervals.
Mean arterial pressure | 24 hours postoperatively
  Mean arterial pressure will be recorded at six predefined intra- and postoperative intervals.
Peripheral Oxygen Saturation | 24 hours postoperatively
  Peripheral Oxygen Saturation will be recorded at six predefined intra- and postoperative intervals.
Stress Level | Two hours postoperatively in the recovery room
  Stress Levels will be measured using the Brief Measure of Emotional Preoperative Stress (B-MEPS) on admission to the operating theatre, at skin suturing, and two hours postoperatively in the recovery room.
  The B-MEPS will be used to assess maternal stress levels. This 12-item tool will be designed as a shorter version of the full Emotional Preoperative Stress scale. It includes items rated on 2-point, 3- point, and 4-point Likert scales, with higher total scores (range 12-36) indicating greater preoperative stress.
Maternal Satisfaction | Two hours postoperatively in the recovery room
  Maternal satisfaction will be evaluated using the Birth Satisfaction Scale-Revised (BSS-R), a widely used and validated instrument in obstetric research. The BSSR comprises 10 items rated on a 5-point Likert scale, ranging from "strongly disagree" [1] to "strongly agree" [5]. Scores will categorize participants into: completely unsatisfied (10-18), unsatisfied (19-26), neutral (27-34), satisfied (35-42), or completely satisfied (43-50).
Apgar score | 5 minutes postoperatively
  Apgar scores will be recorded at 1 and 5 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.